CLINICAL TRIAL: NCT00140413
Title: Endocrine Dysfunction and Growth Hormone Deficiency in Children With Optic Nerve Hypoplasia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Children's Hospital Los Angeles (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Mark Borchert, M.D., Pediatric Neuro-Ophthalmologist, Children's Hospital Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 03.261
Record Dates: First submitted 2005-08-31; First posted 2005-09-01 (Estimated); Results first posted 2015-04-01 (Estimated); Last update posted 2015-04-01 (Estimated); Status verified 2015-03

CONDITIONS: Growth Hormone Deficiency; Septo-Optic Dysplasia; Hypopituitarism
Keywords: Optic Nerve Hypoplasia
MeSH Terms: conditions — Dwarfism, Pituitary; Septo-Optic Dysplasia; Hypopituitarism; Optic Nerve Hypoplasia | interventions — Growth Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment Group 1: Receiving GH Treatment (Experimental): Treatment group assignment was based on subject's stature SDS relative to the mid-parental target height (MPTH) at baseline and subsequent classification as growth deceleration or normal growth. Subjects with growth deceleration were assigned to the GH treatment group in accordance with standard of care. Subjects with normal growth were randomized to treatment or to control (no intervention). The intervention was Nutropin AQ. The starting dose was calculated as 0.3 mg/kg/wk and subsequently modified based on observed length/height velocity and serum IGF-I levels.
  Interventions: Drug: Nutropin AQ
- Treatment Group 2: Control (No Intervention): Treatment group assignment was based on subject's stature SDS relative to the mid-parental target height (MPTH) at baseline and subsequent classification as growth deceleration or normal growth. Subjects with normal growth were randomized to treatment or to control. The control group received no intervention; however, control subjects were switched (crossed over) to the GH replacement group if, during the course of the study, they met criteria for growth deceleration.

INTERVENTIONS:
Drug: Nutropin AQ — Daily injection. Dosage dependent on weight.
  Arms: Treatment Group 1: Receiving GH Treatment

SUMMARY:
Hypotheses:

1. The prevalence of endocrinopathies, and growth hormone (GH) deficiency in particular, among young children diagnosed with optic nerve hypoplasia (ONH) is higher than is commonly thought.
2. Early treatment of children with ONH and GH-deficiency can prevent adverse outcomes.

Aims:

1. Determine the prevalence and types of endocrinopathies in children diagnosed with ONH.
2. Correlate endocrine outcome with radiographic, ocular, and developmental findings in children with ONH.
3. Examine the effect of GH treatment on growth and obesity in children with ONH, GH-deficiency, and either subnormal or normal growth compared to children with ONH that are not GH-deficient.
4. Compare growth outcomes between children with isolated GH-deficiency and those with multiple hormone deficiencies.

DETAILED DESCRIPTION:
Subjects for this study will be recruited from active and newly enrolled subjects in our larger ONH study. The study duration is three years and we anticipate 38 subjects will enroll. Subjects will be recruited for this study if they present with either growth deceleration or at least one subnormal result for IGF-1 or IGFBP-3.

Baseline information collected includes: height, weight, head circumference, examinations by an endocrinologist and ophthalmologist, endocrine laboratory testing, fundus photography, electrophysiology testing, head MRI, and a developmental assessment. A glucagon stimulation test will be performed and subjects who are deemed GH-deficient and who have delayed growth will be assigned to GH treatment, in line with standard clinical practice. Those with normal growth but determined to be GH-deficient by a glucagon stimulation test will be randomized to treatment with GH vs control (no intervention; observation only).

Subjects assigned or randomized to treatment with GH will be provided with GH for the duration of their participation in the study. Enrolled subjects will return every four months to monitor progress. Subjects will undergo a physical examination at each visit, including height, weight, head circumference, and body fat. In addition, subjects assigned or randomized to growth hormone will have laboratory testing of thyroid, IGF-1 and IGFBP-3 hormones, and fasting lipid levels.

ELIGIBILITY:
Inclusion Criteria:

* New subjects diagnosed with ONH less than or equal to 2 years of age and subjects actively enrolled (in currently approved prospective ONH study) will be eligible for enrollment.

Max Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2004-12; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Borchert, MD, Principal Investigator — Childrens Hospital Los Angeles; University of Southern California; Mitchell Geffner, MD, Principal Investigator — Children's Hospital Los Angeles
Locations (1):
- Childrens Hospital Los Angeles, Los Angeles, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from an IRB-approved prospective optic nerve hypoplasia (ONH) registry study at Children's Hospital Los Angeles, between January 2005 through March 2011.
Pre-assignment Details: 39 participants were screened for eligibility: 20 enrolled in the study; 6 failed to meet inclusion criteria; 9 declined participation; and 4 consented to participate but withdrew from the study prior to beginning any study procedures.
Groups:
- Treatment Group 1: Receiving Growth Hormone Treatment: Treatment group assignment was based on subject's stature SDS relative to the mid-parental target height (MPTH) at baseline and subsequent classification as growth deceleration or normal growth. Subjects with growth deceleration were assigned to the GH replacement treatment group in accordance with standard of care. Subjects with normal growth were randomized to treatment or to control (no intervention). The starting dose for GH replacement was calculated as 0.3 mg/kg/wk and subsequently modified based on observed length/height velocity and serum IGF-I levels.
Period: Overall Study
Arm/Group | Treatment Group 1: Receiving Growth Hormone Treatment | Treatment Group 2: Control
Started | 13 | 7
Received at Least One Dose of GH | 13 | 3 (Controls were crossed over to GH if they met criteria for growth deceleration during the study.)
Completed | 10 | 7 (Crossed over subjects were treated as controls for purpose of intent to treat analysis.)
Not Completed | 3 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 2 | 0

BASELINE CHARACTERISTICS:
Population: Please note, 3 children were unenrolled from the study and were therefore excluded from our analysis of results. Therefore, while the participant flow section lists 20 participants, the baseline analysis and results are based on 17 participants.
Groups:
- Treatment Group 1A: Assigned to GH: Subjects with growth deceleration were assigned to the GH replacement treatment group in accordance with standard of care.
- Treatment Group 1B: Randomized to GH: Subjects with normal growth were randomized to GH treatment or to control (no intervention).
- Treatment Group 2: Control: Subjects with normal growth were randomized to treatment or to control (no intervention).
- Total: Total of all reporting groups
Arm/Group | Treatment Group 1A: Assigned to GH | Treatment Group 1B: Randomized to GH | Treatment Group 2: Control | Total
Number analyzed (Participants) | 5 | 5 | 7 | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 5 | 5 | 7 | 17
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Median (Inter-Quartile Range); unit: Months] | 28 [24 to 30] | 41 [33 to 61] | 26 [23 to 50] | 30 [24 to 50]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 4 | 9
  Male | 2 | 3 | 3 | 8
Weight z-score [Median (Inter-Quartile Range); unit: Z-score] — Z-score indicates how many standard deviations an element is from the mean. It is calculated as z = (x - µ) σ, where µ is the mean of the population, and σ is the standard deviation of the population. A positive z-score indicates a datum above the mean, while a negative z-score indicates a datum below the mean. All z-scores were obtained using Epi Info ™ 3.5.4. (Centers for Disease Control, Atlanta, GA).
  Z-score | -1.76 [-2.48 to -1.6] | 0.6 [-0.47 to 1.49] | -1.36 [-1.73 to 0.41] | -1.36 [-1.73 to 0.6]
Stature z-score [Median (Inter-Quartile Range); unit: Z-score] — Z-score indicates how many standard deviations an element is from the mean. It is calculated as z = (x - µ) σ, where µ is the mean of the population, and σ is the standard deviation of the population. A positive z-score indicates a datum above the mean, while a negative z-score indicates a datum below the mean. All z-scores were obtained using Epi Info ™ 3.5.4. (Centers for Disease Control, Atlanta, GA).
  Z-score | -2.16 [-2.35 to -1.94] | -0.95 [-1.73 to -0.22] | -1.3 [-1.79 to -0.91] | -1.73 [-2.16 to -0.95]
Weight-for-stature z-score [Median (Inter-Quartile Range); unit: Z-score] — Weight (wt.) for stature expresses wt. relative to stature (length or height); data are not age specific. The wt. for stature reference data from CDC growth charts compares a child's wt. with the wt. distribution of children of the same stature but not necessarily of the same age.
  Z-score indicates how many standard deviations an element is from the mean. It is calculated as z = (x - µ) σ, where µ is the mean of the population, and σ is the standard deviation of the population. All z-scores were obtained using Epi Info ™ 3.5.4. (Centers for Disease Control, Atlanta, GA).
  Z-score | -0.38 [-0.99 to -0.23] | 1.94 [0.88 to 2.49] | 1.34 [0.22 to 1.73] | 0.82 [-0.38 to 1.91]
Body Mass Index (BMI) z-score [Median (Inter-Quartile Range); unit: Z-score] — BMI adjusts weight for stature and is calculated as weight (kg)/height (m) squared. In children, BMI is age specific. BMI reference data from the CDC growth charts compares a child's BMI with the BMI distribution of children of the same age but not necessarily of the same stature.
  Z-score indicates how many standard deviations an element is from the mean. It is calculated as z = (x - µ) σ, where µ is the mean of the population, and σ is the standard deviation of the population. All z-scores were obtained using Epi Info ™ 3.5.4. (Centers for Disease Control, Atlanta, GA).
  Z-score | -0.2 [-0.5 to 0.11] | 2.06 [1.14 to 2.62] | 1.35 [0.38 to 1.7] | 1.14 [0.05 to 2.06]

OUTCOME MEASURES:

1. Primary Outcome: Change in Anthropometric Measures Over Time
Description: Primary outcome measures included change in stature, weight, BMI, and weight-for-stature z-scores over the course of the study. Z-score indicates how many standard deviations an element is from the mean. It is calculated as z = (x - µ) σ, where µ is the mean of the population, and σ is the standard deviation of the population. A positive z-score indicates a datum above the mean, while a negative z-score indicates a datum below the mean. All z-scores were obtained using Epi Info ™ 3.5.4. (Centers for Disease Control, Atlanta, GA).
Time Frame: Baseline and 36 months
Measure: Median (Inter-Quartile Range); unit: Z-score
Groups:
- Treatment Group 1: Receiving Growth Hormone Treatment: Treatment group assignment was based on subject's stature SDS relative to the mid-parental target height (MPTH) at baseline and subsequent classification as growth deceleration or normal growth. Subjects with growth deceleration were assigned to the GH replacement treatment group in accordance with standard of care. Subjects with normal growth were randomized to treatment or to control (no intervention). The starting daily dose for GH replacement was calculated as 0.3 mg/kg/wk and subsequently modified based on observed length/height velocity and serum IGF-I levels.
- Treatment Group 2: Control: Treatment group assignment was based on subject's stature SDS relative to the mid-parental target height (MPTH) at baseline and subsequent classification as growth deceleration or normal growth. Subjects with normal growth were randomized to treatment or to control. The control group received no intervention; however control subjects were switched (crossed over) to the GH replacement group if, during the course of the study, they met criteria for growth deceleration.
  A total of 7 subjects were randomized to the control group, 3 of whom were crossed over to treatment due to growth deceleration. Outcome measures for these 3 who crossed over were analyzed separately, under Treatment Group 3.
- Treatment Group 3: Control Crossed Over to Treatment: 3 control subjects were switched (crossed over) to the GH replacement group during the course of the study due to growth deceleration.
Arm/Group | Treatment Group 1: Receiving Growth Hormone Treatment | Treatment Group 2: Control | Treatment Group 3: Control Crossed Over to Treatment
Number analyzed (Participants) | 10 | 4 | 3
Z-score
  Change in stature z-score | 1.97 [0.56 to 2.29] | -0.61 [-0.9625 to -0.305] | 1.39 [0.62 to 1.43]
  Change in weight z-score | 1.22 [0.49 to 2.16] | -0.38 [-0.715 to -0.195] | 0.58 [-0.06 to 1.92]
  Change in weight-for-stature z-score | 0.52 [-0.21 to 0.705] | -0.37 [-0.825 to -0.1075] | 0.95 [0.1 to 1.8]
  Change in body mass index (BMI) z-score | -0.06 [-0.24 to 0.39] | -0.505 [-0.7025 to -0.3075] | -1.035 [-1.1525 to -0.9175]

ADVERSE EVENTS:
Time Frame: 36 months (study duration)
Groups:
- Treatment Group 1: Receiving Growth Hormone Treatment: The denominator below (# at risk) is based on the number of subjects in Group 1 who received at least one dose of growth hormone.
- Treatment Group 2: Control: The denominator below (# at risk) is based on the number of subjects in Group 2 who received at least one dose of growth hormone. Per protocol, control subjects received no intervention; however, 3 control subjects were switched (crossed over) to the GH replacement group during the course of the study due to growth deceleration.
Arm/Group | Treatment Group 1: Receiving Growth Hormone Treatment | Treatment Group 2: Control
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/3
Other Adverse Events (participants affected / at risk) | 1/13 | 0/3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Group 1: Receiving Growth Hormone Treatment (N=13) | Treatment Group 2: Control (N=3)
Headache (Nervous system disorders) | 1 (1) | 0 (0) — The event was expected, consistent with the investigator's brochure and reported as a possible risk in the informed consent form.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
With respect to any proposed publication, the PI must submit to the sponsor a copy of the proposed publication at least 2 months prior to submission for the purposes of: providing the sponsor the oppotunity to review and comment on the contents of proposed publication; and to identify any trade secret, proprietary or confidential information to be removed from the proposed publication. The sponsor will provide comments within 30 days of receipt of proposed publication.